## Official title: Polyp Prophylactic Properties of Polyacetylenes in Patients With Previous Polypectomy

Identifier: NCT06335420

Last document update: 07.09.2023

| _ | | | | | | | _ |
|---|---|---|---|---|---|----|---|
| А | D | D | е | n | a | ix | 5 |

**(S1)** 

## Informed Consent for Participation in a Health Science Research Project

**Title of the Research Project**: Polyp Prophylactic Properties of Polyacetylenes in Patients With Previous Polypectomy

## **Declaration by the Participant:**

I have received written and oral information, and I know enough about the purpose, method, benefits, and disadvantages to agree to participate.

I understand that participation is voluntary and that I can withdraw my consent at any time without losing my current or future rights to treatment.

I consent to participate in the research project and have received a copy of this consent form and a copy of the written information about the project for my own use.

| Participant's Name: | |
|---|---|
| Date: | Signature: |
| Would you like to be info you?: | ormed about the results of the research project and any potential consequences for |
| Yes (tick) No | (tick) |
| Declaration by the Infor | mer: |
| I declare that the partici | pant has received oral and written information about the study. |
| To the best of my knowl in the study. | edge, sufficient information has been provided to make a decision about participation |
| Name of the Informer: _ | |
| Date: | Signature: |

Registration Number Scientific Ethics Committee: 105989 / 07.09.2023